CLINICAL TRIAL: NCT03683654
Title: Mining the Urinary and Serum Metabolome for Discovery of Novel Biomarkers of Dietary Exposure in the EPIC Calibration Study
Brief Title: Discovery of Novel Biomarkers of Dietary Exposure in the EPIC Calibration Study
Status: Completed | Type: Observational
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Imperial College London (Other); Centre for Research in Epidemiology and Population Health (CESP) (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); German Cancer Research Center (Other); German Institute of Human Nutrition (Other); Hellenic Health Foundation (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Cancer Prevention and Research Institute, Italy (Other); Federico II University (Other); Center for Cancer Prevention (CPO) (Unknown); Azienda Sanitaria Provinciale Ragusa (Other)
Responsible Party: Sponsor
Other Study IDs: PP201204-12
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Dietary Exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 24-hour urine samples Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Identify Biomarkers of Dietary Intake in Healthy Subjects — Observational study. No intervention.

SUMMARY:
This proposal aims at identifying new biomarkers of dietary exposure using metabolomic approaches. This project is based on the European Prospective Investigation on Cancer and Nutrition (EPIC) Calibration Study and more particularly upon a subset of 494 men and women from 4 European countries (Germany, Greece, Italy and France). Urine and blood samples are analyzed by untargeted metabolomics.

DETAILED DESCRIPTION:
Subjects participating in the study are characterized by the availability of one 24-hr urine sample, blood serum, 24-hr dietary recall (24HDR) and food frequency questionnaire (FFQ) data.

The main objectives of the proposal are:

1. To collect a set of high-quality metabolomic data containing rich information on the food-derived metabolome.
2. To mine this data in different Metabolome-Wide Association Studies in order to identify food-derived metabolites discriminating consumers and non-consumers of various foods, nutrients and dietary patterns.
3. To identify the food-derived metabolites characteristic of the consumption of the different foods/nutrients and dietary patterns.

ELIGIBILITY:
Inclusion criteria:

* Aged 30-70
* Healthy
* Residing within Europe.
* Have donated one 24-hr urine sample, blood serum.
* Have filled one 24-hr dietary recall (24HDR) and food frequency questionnaire (FFQ).

Exclusion criteria:

* 24-hr urine sample and 24-hr dietary recall not collected on a same day.
* Incomplete collection of 24-hr urine sample.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 494 men and women from 4 European countries (Germany, Greece, Italy and France) selected from the EPIC Calibration study. Different settings by centre; mostly general population with some exceptions: women of a health insurance company for teachers and school workers (France), women attending breast cancer screening (Florence-Italy), mainly blood donors (most centers in Italy) and a cohort consisting predominantly of vegetarians (the 'health-conscious' group in Oxford, UK).
Sampling Method: Non-Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2012-04-26 (Actual); Primary Completion 2013-02-23 (Actual); Study Completion 2013-02-23 (Actual)

PRIMARY OUTCOMES:
Metabolite concentrations in plasma and urine | 1 day
  Food-derived Metabolite concentrations in plasma and urine are measured by high resolution mass spectrometry coupled to ultrahigh performance chromatography.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Riboli E, Hunt KJ, Slimani N, Ferrari P, Norat T, Fahey M, Charrondiere UR, Hemon B, Casagrande C, Vignat J, Overvad K, Tjonneland A, Clavel-Chapelon F, Thiebaut A, Wahrendorf J, Boeing H, Trichopoulos D, Trichopoulou A, Vineis P, Palli D, Bueno-De-Mesquita HB, Peeters PH, Lund E, Engeset D, Gonzalez CA, Barricarte A, Berglund G, Hallmans G, Day NE, Key TJ, Kaaks R, Saracci R. European Prospective Investigation into Cancer and Nutrition (EPIC): study populations and data collection. Public Health Nutr. 2002 Dec;5(6B):1113-24. doi: 10.1079/PHN2002394. PMID 12639222
- [Background] Slimani N, Ferrari P, Ocke M, Welch A, Boeing H, Liere M, Pala V, Amiano P, Lagiou A, Mattisson I, Stripp C, Engeset D, Charrondiere R, Buzzard M, Staveren W, Riboli E. Standardization of the 24-hour diet recall calibration method used in the european prospective investigation into cancer and nutrition (EPIC): general concepts and preliminary results. Eur J Clin Nutr. 2000 Dec;54(12):900-17. doi: 10.1038/sj.ejcn.1601107. PMID 11114689
- [Result] Edmands WM, Ferrari P, Rothwell JA, Rinaldi S, Slimani N, Barupal DK, Biessy C, Jenab M, Clavel-Chapelon F, Fagherazzi G, Boutron-Ruault MC, Katzke VA, Kuhn T, Boeing H, Trichopoulou A, Lagiou P, Trichopoulos D, Palli D, Grioni S, Tumino R, Vineis P, Mattiello A, Romieu I, Scalbert A. Polyphenol metabolome in human urine and its association with intake of polyphenol-rich foods across European countries. Am J Clin Nutr. 2015 Oct;102(4):905-13. doi: 10.3945/ajcn.114.101881. Epub 2015 Aug 12. PMID 26269369
- See also: Website of the EPIC cohort study — http://epic.iarc.fr/